CLINICAL TRIAL: NCT05452057
Title: Prehabilitation for Adult Spinal Deformity Surgery: a Feasibility Randomized Controlled Trial
Brief Title: Prehab for Adult Spinal Deformity Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Daniel Santa Mina, Clinician Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-5303
Record Dates: First submitted 2022-06-30; First posted 2022-07-11 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Spinal Deformity
Keywords: Prehabilitation; Exercise; Stress management; Nutrition
MeSH Terms: conditions — Motor Activity | interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: Randomized (1:1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): This will include an individualized, light to moderate intensity resistance training and aerobic exercise components. Each prescribed session will include: a minute warm-up, aerobic exercise, resistance training, and a cool-down, but may be modified to accommodate the participants exercise ability.
  A registered dietitian will provide an individualized nutrition assessment and counselling session within the first week of prehabilitation and again in the week prior to surgery.
  A staff psychologist or psychology resident will deliver a ~60-minute psychoeducation session that focuses on stress management via relaxation, mindfulness, goal setting, and strategies to overcoming barriers to practice. In the week prior to surgery, participants will be offered a second consultation with the psychology team member to review their stress management experiences and provide further support for the acute perioperative period.
  Interventions: Behavioral: Prehabilitation
- Usual care (No Intervention): Usual care group will be asked to resume your typical lifestyle behaviours until the date of the surgery and will be provided with publicly available resources on physical activity, diet, and stress management.

INTERVENTIONS:
Behavioral: Prehabilitation — A Registered Kinesiologist will provide your exercise prescription during your first visit for the study. Your exercise sessions will consist of moderate-intensity cardiovascular (or aerobic) exercise, like brisk walking, for 30 minutes. You will also perform resistance exercises (weight lifting) for 30 minutes that will help strengthen your muscles with a focus on muscles that may be affected by your surgery. To complete your exercises, you will receive resistance bands, exercise ball, and exercise manual.
  You will also meet with a Registered Dietician within a week of consent to receive information on healthy eating and you will receive protein to improve your nutritional health.
  A consult with an expert in psychology to discuss ways to reduce your stress within a week of consent. Some strategies to help reduce your stress may include breathing exercises, being mindful, or other relaxation methods.
  Arms: Prehabilitation

SUMMARY:
Prehabilitation is defined as the process of enhancing patients' functional capacity and overall fitness to enable them to withstand a forthcoming stressor (e.g. surgery). Although there are different models of prehabilitation, multimodal prehabilitation is recommended to address the physical and psychological health outcomes prior to surgery. Multimodal prehabilitation commonly consists of exercise-training, nutritional, and psychological support. Evidence suggests that prehabilitation improves preoperative physical fitness and reduces postoperative complications and length of stay in patients undergoing major abdominal surgery. However, the evidence for the feasibility and effects in spinal deformity surgery are less understood. This study is a two arm, pilot randomized controlled trial to assess the feasibility of a multimodal prehabilitation program prior to surgery for spinal deformity in adults. Participant outcomes will be measured using standardized fitness testing, self-report questionnaires, and medical record reviews at baseline, one week preoperatively, and at 30 days postoperatively.

DETAILED DESCRIPTION:
Spinal deformity is defined as a curvature in the spine where the alignment is outside of defined normal limits in the sagittal (e.g., kyphosis, lordosis), or coronal plane (e.g., scoliosis). The severity of symptoms among patients with spinal deformity varies and is contingent upon the type and extent of deformity. Studies have shown that adult patients with symptomatic spinal deformity have similar or worse patient-reported health-related quality of life (HRQOL) compared with other pathological conditions such as arthritis, chronic pulmonary disease, congestive heart failure, diabetes, and cancer. Over the last decade, multiple studies have demonstrated a significant improvement in patient HRQOL, disability and leg pain following spinal deformity surgery at 2-years of follow up. In contrast, patients who are treated non-surgically do not exhibit significant HRQOL changes compared to baseline. Spinal deformity surgery, however, can be associated with complications, with rates as high as 77%. Possible complications include hemorrhage, cerebrospinal fluid leak, screw malposition, ischemic optic neuropathy, thromboembolic events, cardiopulmonary complications, and infection. Recovery from surgery is long-term and challenging, with an expectation that patients may feel worse for up to 3 months after surgery. Moreover, length of hospital stay (LOS), discharge to inpatient rehabilitation, and additional post-discharge, home-care support following spinal deformity surgery are significant drivers of health care costs. In fact, LOS has been reported up to 100 days, with predictors of increased LOS including frailty and functional status. Thus, strategies that can improve preoperative functional status, and subsequently reduce postoperative LOS and improve postoperative recovery trajectories are important for adults undergoing surgery for spinal deformity.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for spinal deformity surgery;
* recruited at least 12 weeks preoperatively;
* a frailty score of 0.27 or greater as indicated by the Modified Frailty index-11; and
* proficient in English to comprehend informed consent and intervention instructions

Exclusion Criteria:

* Refusal to be randomized;
* have significant comorbidity precluding participation in prehabilitation exercises (including Canadian Cardiovascular Society class III/IV coronary disease; New York Heart Association class III/IV congestive heart failure; neurological or musculoskeletal disorder prohibiting exercise; major neuropsychiatric disorder)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility assessment: Recruitment and Enrollment | 6 months
  - Recruitment success will be measured by the proportion of participants who are randomized divided by the number of identified eligible patients. Reasons for non-participation will be collected. The feasibility target is 25%.
Feasibility assessment: Intervention fidelity | pre-operative
  - Reasons for, all or part, the intervention not being delivered as intended will be recorded. The kinesiologist will communicate with prehabilitation participants via telephone and/or email weekly to ensure program compliance, record adherence, support appropriate progression, and to address any barriers to exercise that may prevent participation.
Feasibility assessment: Adherence, | pre-operative
  - Adherence to stress management and utilization of smoking cessation tools (as required) will be recorded weekly using a logbook within the participant manuals. This includes the attendance to consultations with RD and psychologist, number of relaxation sessions per week; compliance with RD recommendations for dietary behaviours, protein supplementation, and for smokers, the tools used, and the number of times accessed.
Feasibility assessment: Retention | 6 months
  - The frequency of drop-out during program participation will be documented including reasons for drop-out. The feasibility target for attrition is less than 15%.
Feasibility assessment: Safety and adverse events | 6 months
  - Any safety or adverse events related to the prehabilitation intervention will be reported during weekly telephone calls with participants. Reporting and grading will follow the Common Terminology Criteria for Adverse Events version 5.0.
Feasibility assessment: Cost. | 6 months
  - Cost of delivery for the prehabilitation intervention will be captured based on the individual perspective. This will be calculated based on the quantity of resources consumed, the unit cost of those resources related to the intervention, and personnel cost for delivery of the intervention.

SECONDARY OUTCOMES:
Clinical outcomes: hospital length of stay | Post-operative
  - Postoperative LOS will be recorded from the participant medical record in days from the time of surgery until hospital discharge.
Clinical outcomes: Discharge disposition | Post-operative
  Discharge destination (i.e. rehabilitation) and total inpatient stay (if applicable) will recorded in days.
Clinical outcomes: Complications | 6 months
  Complications, including mortality, will follow the Clavien-Dindo classification. Any health event that requires readmission will also be documented. This will be recorded during hospitalization and within 6 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Santa Mina, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada